CLINICAL TRIAL: NCT02293681
Title: A Multicenter and Observational Study to Assess the Effectiveness of Infliximab Comparing With Conventional Therapy in Ankylosing Spondylitis Subjects With Hip Involvement
Brief Title: An Observational Study of Infliximab in Participants Suffering From Ankylosing Spondylitis With Hip Involvement
Acronym: RECOVERY
Status: Terminated | Type: Observational
Why Stopped: The project was stopped by 31-May-2017 because of internal owner decision from out of balance enrollment from two groups.
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR104999; REMICADEAKS4006 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2014-11-14; First posted 2014-11-18 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Spondylitis, Ankylosing
Keywords: Spondylitis, Ankylosing; Infliximab; Non-steroidal anti-inflammatory drugs; Disease-modifying anti-rheumatic drugs
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Infliximab; Anti-Inflammatory Agents, Non-Steroidal; Antirheumatic Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 52 Weeks
Biospecimen Retention: Samples Without DNA — Blood samples will be retained for the assessment of laboratory parameters: CRP = C-reactive protein; ESR = erythrocyte sedimentation rate.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Infliximab and/or NSAIDs and DMRADs: Participants receiving intravenous infusion of infliximab with or without non-steroidal anti-inflammatory drugs (NSAIDs: aspirin, ibuprofen and naproxen) and Disease-modifying anti-rheumatic drugs (DMRADs: methotrexate (MTX), sulfasalazine, and thalidomide) will be observed.
  Interventions: Drug: Infliximab; Drug: NSAIDs; Drug: DMARDs
- Cohort 2: NSAIDs and DMARDs: Participants receiving NSAIDs (aspirin, ibuprofen and naproxen) and DMARDs (MTX, sulfasalazine, and thalidomide) will be observed.
  Interventions: Drug: NSAIDs; Drug: DMARDs

INTERVENTIONS:
Drug: Infliximab — This is an observational study. Participants receiving intravenous infusion of infliximab will be observed.
  Groups: Cohort 1: Infliximab and/or NSAIDs and DMRADs
Drug: NSAIDs — This is an observational study. Participants receiving aspirin, ibuprofen and naproxen as NSAIDs will be observed.
Drug: DMARDs — This is an observational study. Participants receiving methotrexate (MTX), sulfasalazine, and thalidomide as DMRADs will be observed.

SUMMARY:
The purpose of this observational (a study that follows participants forward in time) study is to compare the functional improvement of hip joint using Harris hip score between 2 treatment groups (infliximab and conventional therapy) at Week 30 in ankylosing spondylitis (an autoimmune disease causing chronic inflammation at tendon ends and ligament attachment points) participants with hip involvement.

DETAILED DESCRIPTION:
This is a multi-center (when more than 1 hospital or medical school team work on a medical research study), observational study to compare the effectiveness of infliximab with conventional therapies in ankylosing spondylitis participants with hip joint involvement. The study will be conducted in 3 parts: a 14-day screening, a 30-week first follow-up (Follow-up 1), and an additional 22-week follow-up (Follow-up 2) up to Week 52. Participants will be assigned to two groups based on the current treatments they are receiving: cohort 1 participants receiving infliximab with or without combination of disease modifying drugs (DMARDs-such as Sulfasalazine, Methotrexate and Thalidomide) and/or non-steroidal anti-inflammatory drugs (NSAIDs) and in cohort 2 who are receiving DMARDs and/or NSAIDs for treatment of pain will be observed. Participants will primarily be assessed for change in harris hip score. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with ankylosing spondylitis (AS) (according to the modified New York Criteria for AS) at least 3 months prior to the Day 1 in the Follow-up I phase with symptoms of active disease atScreening/Baseline
* Hip pain and duration of hip symptom less than 2 years
* Harris hip score less than (<) 70
* Hip involvement proven by Magnetic resonance imaging (MRI)
* Being treated with infliximab and conventional therapy for 2 weeks to 6 months

Exclusion Criteria:

* Participant has a history of hip joint disability which was considered irreversible
* Participant has a history of hip joint replacement
* Participant has a history of treatment with biologics other than infliximab less than 6 months prior to study entry

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants suffering from ankylosing spondylitis with hip involvement.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2015-04-10 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Harris Hip Score at Week 30 | Baseline and Week 30
  Harris hip score, a physician-assessed scoring method consisting of 10 items: pain, limp, support, distance walked, sitting, enter public transportation, stairs, put on shoes and socks, absence of deformity and range of motion. The scoring system covers domains like pain, function, absence of deformity and range of motion. The total Harris hip score has a maximum of 100 points with a higher score indicating a better hip function: Excellent (90-100), Good (80-89), Fair (70-79) and Poor (<70).

SECONDARY OUTCOMES:
Change From Baseline in Bath Ankylosing Spondylitis Disease Activities Index (BASDAI) Score at Week 30 and 52 | Baseline, Week 30 and 52
  The BASDAI is used to measure the ankylosing spondylitis (AS) disease severity. It consists of 6 questions: fatigue, spinal pain, arthralgia (joint pain) or swelling, enthesitis (inflammation of tendons and ligaments), and morning stiffness (2 questions: duration and severity). Each question is an easy to answer 10cm visual analog scale (VAS), with 1 being none, and 10 being very severe. In order to give each of the 5 symptoms equal weight, the mean of the 2 questions about morning stiffness will be added to the total of the remaining 4 scores, and the final BASDAI score (ranging 0-10) is the average of the overall total score. Higher BASDAI score indicates more severe AS symptom.
Change From Baseline in Bath Ankylosing Spondylitis Functional Index (BASFI) Score at Week 30 and 52 | Baseline, Week 30 and 52
  The BASFI is composed with 10 questions to assess the disease severity, including the first 8 questions regarding to functional anatomy related activities and the remaining 2 questions related to daily activities of AS participants. Each question is a 10cm VAS with a value between 0 (easy) and 10 (impossible). The final BASFI score is the mean of the 10 scores. Higher BASFI score indicates more severe functional limitations of the participant due to AS.
Change From Baseline in Bath Ankylosing Spondylitis Metrology Index (BASMI) Score at Week 30 and 52 | Baseline, Week 30 and 52
  The BASMI is an accurate and reproducible metrology index developed to assess the clinical changes in spinal movements of AS participants. This index consists of 5 clinical measurements, including lumber side flexion, tragus to wall, lumbar flexion (modified Schober's), intermalleoar distance and cervical rotation. The potential scores for each measurement are 0, 1, and 2, indicating a disease severity of mild, moderate and severe, respectively. A higher BASMI score indicates a more severe movement limitation due to AS.
Change From Baseline in Ankylosing Spondylitis Disease Activity Score (ASDAS) at Week 30 and 52 | Baseline, Week 30 and 52
  The ASDAS is composite score based on the calculation of 5 disease activities: 4 are participant's reported outcomes (back pain, duration of morning stiffness, participant global and peripheral pain/swelling) and one serologic inflammation marker (creatinine reactive protein - CRP). The score is the sum of the 5 items with different specified weights, with a minimum of 0 and no upper limit. Thus this index can reflect both long term disease activity and acute phase status. There are 3 cut-offs in score to show: a) the 4 states of disease activity: inactive disease (<1.3), moderate disease activity (1.3-2.1), high disease activity (2.1-3.5) and very high disease activity (>3.5). b) effectiveness of the treatment, two validated cut-offs were developed: a change of 1.1-2.0 (clinically important improvement) and a change >2.0 (major improvement).
Change From Baseline in Harris Hip Score at Week 14 and 52 | Baseline, Week 14 and 52
  Harris hip score, a physician-assessed scoring method consisting of 10 items: pain, limp, support, distance walked, sitting, enter public transportation, stairs, put on shoes and socks, absence of deformity and range of motion. The scoring system covers domains like pain, function, absence of deformity and range of motion. The total Harris hip score has a maximum of 100 points with a higher score indicating a better hip function: Excellent (90-100), Good (80-89), Fair (70-79) and Poor (<70).
Assessment of Improvement in Hip Joint | Baseline, Week 30 and 52
  Radiological improvements of hip joint will be assessed using magnetic resonance imaging (MRI) and X-ray examinations.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (6):
- China (6):
  - Beijing
  - Changsha
  - Chengdu
  - Guangzhou
  - Shanghai
  - Xi'an